CLINICAL TRIAL: NCT05480735
Title: EffectiveNess of a Multimodal preHAbilitation Program in patieNts With Bladder canCEr Undergoing Cystectomy. The ENHANCE Randomized Controlled Trial
Brief Title: EffectiveNess of a Multimodal preHAbilitation Program in patieNts With Bladder canCEr Undergoing Cystectomy
Acronym: ENHANCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: UMC Utrecht (Other); University Medical Center Groningen (Other); Radboud University Medical Center (Other); Rijnstate Hospital (Other); Noordwest Ziekenhuisgroep (Other); Erasmus Medical Center (Other); Maastricht University Medical Center (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL78792.031.22
Record Dates: First submitted 2022-07-14; First posted 2022-07-29 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Bladder Carcinoma
Keywords: prehabilitation; bladder cancer; exercise; smoking cessation; nutritional support; surgical complications; cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Motor Activity; Smoking Cessation | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation group (Experimental): The intervention group will participate in a prehabilitation program of approximately 4-6 weeks before surgery, and additionally during neoadjuvant chemotherapy if applicable. The program consist of a tailored exercise program, nutritional support and if relevant smoking cessation and/or psychological counselling. The exercise program is under supervision of an oncology specialized physiotherapist and comprises aerobic-, resistance- and breathing- and relaxation exercises. A dietician will provide nutritional support and give dietary advice to increase protein intake, including a supplement containing 30 g of whey-protein daily and after supervised training. Patients who score high on anxiety and depression will be offered a referral to a psychologist. Intensive counselling and nicotine replacement therapy will be offered to all patients who smoke.
  Patients will be asked to keep a diary to track unsupervised activity and to track intake of the protein supplementation.
  Interventions: Behavioral: Prehabilitation
- Control group (No Intervention): Patients randomized to the control group will receive care as usual according to local ERAS guideline implementation. In addition, they will receive a leaflet with the recent guidelines regarding physical activity, dietary advice, and smoking cessation. Their actual physical activity level will be obtained via questionnaire.

INTERVENTIONS:
Behavioral: Prehabilitation — Multimodal prehabilitation program
  Arms: Prehabilitation group

SUMMARY:
Currently, the potential value of a multimodal prehabilitation program in bladder cancer has not been extensively studied. The investigators designed the ENHANCE study to assess the effect of a structured multimodal prehabilitation program in 154 patients with bladder cancer on the number (primary endpoint) and severity of complications within 90 days, length of hospital stay, readmissions, physical fitness, muscle strength, physical functioning, nutritional status, smoking behaviour, anxiety and depression, fatigue, quality of life, physical activity, tumor tissue characteristics, and healthcare costs.

DETAILED DESCRIPTION:
The ENHANCE study is a multicenter, randomized controlled trial. The intervention group will participate in a prehabilitation program of 4-6 weeks before surgery, and additionally during neoadjuvant chemotherapy if applicable. The prehabilitation program consist of a tailored exercise program, nutritional support and if relevant smoking cessation and/or psychological counselling. The exercise program is under supervision of an oncology specialized physiotherapist and comprises aerobic-, resistance- and breathing- and relaxation exercises. Patients will be asked to be physically active for an additional 2 times a week for at least 30 minutes. A dietician will provide nutritional support and give dietary advice to increase protein intake to enhance the anabolic effect on muscle mass. Additionally, patients will receive a supplement containing 30 g of high quality whey-protein daily preferably before sleep and after the supervised training. Patients who score high on anxiety and depression will be offered a referral to a psychological support. Intensive counselling and nicotine replacement therapy will be offered to all patients who smoke. Patients in the intervention group will be asked to keep a diary to track unsupervised activity and to track intake of the protein supplementation. The physical activity level in both groups will be obtained via questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, primary, bladder cancer (cTa-4N0/N+M0),
* Planned to undergo radical cystectomy,
* Age ≥ 18 years.

Exclusion Criteria:

* Subjects with severe cognitive or psychiatric disorders,
* Subjects who are operated within 3 weeks,
* Subjects with insufficient command of the Dutch language, which precludes them from following study instructions or completing study questionnaires,
* Subjects who have contraindications to safely perform exercise training or testing (i.e., CPET),
* Subject who are unable or unwilling to participate in the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Complications | 0-12 weeks post-surgery (measured 4 weeks and 12 weeks post-surgery)
  The proportion of patients having Clavien-Dindo grade 2 or higher perioperative complications; obtained from the medical records

SECONDARY OUTCOMES:
High grade complications | 0-12 weeks post-surgery
  Clavien Dindo grade 3 or higher
Duration of hospital stay | 0-12 weeks post-surgery
  Time from admission until hospital discharge
Readmissions | 0-12 weeks post-surgery
  Hospital readmission as recorded in medical file
Disease status | 0-12 weeks post-surgery
  Progression/recurrence, any additional treatment as recorded in medical file
Change in cardiorespiratory fitness | T0a (baseline), T1 (within 1 week before surgery)
  Assessed via cardiopulmonary exercise test (CPET)
Change in muscle strength | T0a (baseline), T1 (within 1 week before surgery), T3 (12 weeks post-surgery)
  Grip strength
Change in muscle strength | T0a (baseline), T1 (within 1 week before surgery), T3 (12 weeks post-surgery)
  30s chair stands
Change in physical performance | T0a (baseline), T1 (within 1 week before surgery), T3 (12 weeks post-surgery)
  Short Physical Performance Battery (SPPB)
Change in nutritional status | T0a (baseline), T1 (within 1 week before surgery), T3 (12 weeks post-surgery)
  Short Form- Patient Generated Subjective Global Assessment (SF-PGSA)
Change in body composition | T0a (baseline), T1 (within 1 week before surgery), T3 (12 weeks post-surgery)
  Fat free mass and fat mass assessed by Scale Bioelectrical Impedance Analysis (BIA)
Nil per mouth consumption during hospitalization | 0-12 weeks post-surgery
  The total days as recorded in medical file
Change in weight | T0a (baseline), T1 (within 1 week before surgery), T3 (12 weeks post-surgery)
  Measured in KG
Height | T0a (baseline) - T3 (12 weeks post-surgery)
  Measured in cm
Change in smoking status | T0a (baseline), T0b (if applicable: after neoadjuvant chemotherapy), T1 (within 1 week before surgery), T2 (4 weeks post-surgery), T3 (12 weeks post-surgery)
  Self-developed questionnaire
Sense of coherence (SOC) | T0a (baseline)
  13-item SOC questionnaire
Change in fatigue | T0a (baseline), T0b (if applicable: after neoadjuvant chemotherapy), T1 (within 1 week before surgery), T2 (4 weeks post-surgery), T3 (12 weeks post-surgery)
  MFI questionnaire
Change in HRQoL | T0a (baseline), T0b (if applicable: after neoadjuvant chemotherapy), T1 (within 1 week before surgery), T2 (4 weeks post-surgery), T3 (12 weeks post-surgery)
  EORTC QLQ-C30
Change in muscle invasive bladder cancer specific scores | T0a (baseline), T0b (if applicable: after neoadjuvant chemotherapy), T1 (within 1 week before surgery), T2 (4 weeks post-surgery), T3 (12 weeks post-surgery)
  EORTC QLQ-BLM30
Change in health status | T0a (baseline), T0b (if applicable: after neoadjuvant chemotherapy), T1 (within 1 week before surgery), T2 (4 weeks post-surgery), T3 (12 weeks post-surgery)
  EQ-5D-5L
Change in physical activity | T0a (baseline), T0b (if applicable: after neoadjuvant chemotherapy), T1 (within 1 week before surgery), T2 (4 weeks post-surgery), T3 (12 weeks post-surgery)
  SQUASH questionnaire
Change in anxiety and depression | T0a (baseline), T0b (if applicable: after neoadjuvant chemotherapy), T1 (within 1 week before surgery), T2 (4 weeks post-surgery), T3 (12 weeks post-surgery)
  HADS questionnaire
Intervention costs | T0a (baseline) - T3 (12 weeks post-surgery)
  Cost analysis
Healthcare resources consumption | T0a (baseline) - T3 (12 weeks post-surgery) (measured within 1 week before surgery, 4 and 12 weeks post-surgery and if applicable : after neoadjuvant chemotherapy)
  Medical Consumption Questionnaire (iMCQ)
Work status | T0a (baseline) - T3 (12 weeks post-surgery)
  Productivity Cost Questionnaire (iPCQ)
Satisfaction with prehabilitation in intervention group and evaluation in control group | T3 (12 weeks post-surgery)
  Self-developed questionnaire
Non participation analysis | T0a (baseline)
  Identify clinical and sociodemographic variables that are related to non-participation of patients in this trial via questionnaire
Hypoxia | T3 (12 weeks post-surgery)
  To study the effectiveness of the prehabilitation program in terms of inducing favorable changes in tumor hypoxia markers

OTHER OUTCOMES:
Overall and bladder-cancer specific survival | 0-60 months
  Exploratory outcome
Progression-free survival | 0-60 months
  Exploratory outcome

CONTACTS AND LOCATIONS:
Locations (8):
- Netherlands (8):
  - Erasmus Medical Center, Rotterdam, Doctor Molewaterplein 40
  - Radboudumc, Nijmegen, Geert Grooteplein Zuid 10
  - UMC Groningen, Groningen, Hanzeplein 1
  - UMC Utrecht, Utrecht, Heidelberglaan 100
  - Catharina Ziekenhuis, Eindhoven, Michelangelolaan 2
  - Maastricht UMC+, Maastricht, P. Debyelaan 25
  - Rijnstate, Arnhem, Wagnerlaan 55
  - Noordwest Ziekenhuisgroep, Alkmaar, Wilhelminalaan 12

IPD SHARING:
Plan to Share IPD: Undecided
Patients are asked informed consent for data sharing with POLARIS consortium

REFERENCES:
- [Derived] Akdemir E, Sweegers MG, Vrieling A, Rundqvist H, Meijer RP, Leliveld-Kors AM, van der Heijden AG, Rutten VC, Koldewijn EL, Bos SD, Wijburg CJ, Marcelissen TAT, Bongers BC, Retel VP, van Harten WH, May AM, Groen WG, Stuiver MM. EffectiveNess of a multimodal preHAbilitation program in patieNts with bladder canCEr undergoing radical cystectomy: protocol of the ENHANCE multicentre randomised controlled trial. BMJ Open. 2023 Mar 7;13(3):e071304. doi: 10.1136/bmjopen-2022-071304. PMID 36882246